CLINICAL TRIAL: NCT00690638
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate Safety and Efficacy of PHX1149T as Monotherapy in Subjects With Type 2 Diabetes Mellitus
Brief Title: Safety and Efficacy Study of Dutogliptin/PHX1149T to Treat Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Phenomix (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Hans-Peter Guler, MD / Chief Medical Officer, Phenomix Corporation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHX1149-PROT301; EudraCT 2008-002614-22
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: dutogliptin; PHX1149; DPP4 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dutogliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Experimental): PHX1149T 200 mg
  Interventions: Drug: PHX1149T
- 3 (Experimental): PHX1149T 400 mg
  Interventions: Drug: PHX1149T

INTERVENTIONS:
Drug: PHX1149T — 200 mg
  Other Names: dutogliptin
  Arms: 2
Drug: PHX1149T — 400 mg
  Other Names: dutogliptin
  Arms: 3
Drug: Placebo — Placebo
  Arms: 1

SUMMARY:
A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate Safety and Efficacy of PHX1149T as Monotherapy in Subjects with Type 2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, drug naïve or willing to wash-out from existing oral therapy
* BMI 25 to 48 kg/m2, inclusive
* HbA1c 7.0% - 10.0%, inclusive
* Age 18 to 75 years, inclusive

Exclusion Criteria:

* Currently on 3 or more oral antidiabetic drugs or insulin.
* Type 1 diabetes mellitus

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To demonstrate changes in HbA1c | Day 28 to Day 196

CONTACTS AND LOCATIONS:
Locations (62):
- United States (13):
  - Norwalk, California
  - Orange, California
  - Santa Ana, California
  - Daytona Beach, Florida
  - Kissimmee, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Brockton, Massachusetts
  - St Louis, Missouri
  - Cincinnati, Ohio
  - El Paso, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
- Argentina (7):
  - Caba, Buenos Aires
  - La Plata, Buenos Aires
  - Lanús, Buenos Aires
  - Paraná, Entre Ríos Province
  - Salta, Salta Province
  - Rosario, Santa Fe Province
  - Corrientes
- India (9):
  - Hyderabad, Andhara Pradesh
  - Bangalore, Karnataka
  - Kalaburagi, Karnataka
  - Mumbai, Maharashtra
  - Nagpur, Maharashtra
  - Nashik, Maharashtra
  - Navi Mumbai, Maharashtra
  - Pune, Maharashtra
  - Chennai, Tamil Nadu
- Malaysia (4):
  - Kelantan
  - Kuala Lumpur
  - Perak
  - Sarawak
- Peru (6):
  - Arequipa, Arequipa
  - Chiclayo-Lambayeque, Chiclayo
  - Lima Cercado, Lima region
  - Lince, Lima region
  - San Miguel, Lima region
  - San Isisdro, Lima
- Philippines (4):
  - Manila, NCR
  - Quezon City, NCR
  - San Juan City, NCR
  - Cebu City, VII
- Romania (7):
  - Brasov, Brașov County
  - Jud. Brasov, Brașov County
  - Sector 1, Bucharest
  - Sector 2, Bucharest
  - Galati, Galați County
  - Ploieşti, Ploiesti
  - Sibiu, Sibiu County
- Thailand (2):
  - Ratchatavi, Bangkok
  - Muang, Changwat Khon Kaen
- Ukraine (10):
  - Simferopol, Crimean Autonomy Republic
  - Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Kharkiv, Kharkivs’ka Oblast’
  - 2A Postysheva Pr., Kharkov
  - Kiev, Kyiv City
  - Kyiv, Kyiv Oblast
  - Lviv, Lviv Oblast
  - Poltava, Poltava Oblast
  - Vinnytsa, Vinnytsa
  - Zaporizhzhia, Zaporizhzhia Oblast